CLINICAL TRIAL: NCT07187258
Title: the Use of Tranexamic Acid in Preventing Intraoperative and Postoperative Hemorrahge in Bariatric Surgery
Brief Title: the Use of Tranexamic Acid to Prevent the Bleeding in Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elshwadfy Nageeb, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-204-2024
Record Dates: First submitted 2025-08-23; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Haemorrhage; Bariatric Surgery Candidate
Keywords: bleeding - sleeve gastrectomy (SG)
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1 ratio to receive tranexamic acid or placebo using a computer-generated block randomization sequence (block size = 4) prepared by an independent pharmacist. Allocation concealment was maintained with sequentially numbered, opaque, sealed envelopes. The pharmacist also prepared indistinguishable infusion bags containing either tranexamic acid (1 g diluted in 100 mL of 0.9% saline) or placebo (100 mL of 0.9% saline). The infusion was administered intravenously over 10-15 minutes immediately after induction of anesthesia and before skin incision, at a maximum rate of 100 mg per minute. Blinding was maintained for patients, anesthesiologists, scrub nurses, and all postoperative assessors, while the operating surgeon was necessarily unblinded, becoming aware of allocation only once the envelope was opened in the operating room. All analyses were performed according to the intention-to-treat principle.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were randomized in a 1:1 ratio to receive tranexamic acid or placebo using a computer-generated block randomization sequence (block size = 4) prepared by an independent pharmacist. Allocation concealment was maintained with sequentially numbered, opaque, sealed envelopes. The pharmacist also prepared indistinguishable infusion bags containing either tranexamic acid (1 g diluted in 100 mL of 0.9% saline) or placebo (100 mL of 0.9% saline). The infusion was administered intravenously over 10-15 minutes immediately after induction of anesthesia and before skin incision, at a maximum rate of 100 mg per minute. Blinding was maintained for patients, anesthesiologists, scrub nurses, and all postoperative assessors, while the operating surgeon was necessarily unblinded, becoming aware of allocation only once the envelope was opened in the operating room. All analyses were performed according to the intention-to-treat principle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic acid (1 g diluted in 100 mL of 0.9% saline (Experimental): TXA 1gm dilutedin 100 ml of .9% normal saline Will be given as IV infusion Before anasthesia
  Interventions: Drug: tranexamic acid (1 g diluted in 100 mL of 0.9% saline
- placebo (100 mL of 0.9% saline). (Placebo Comparator): Placebo diluted in 100 ml of .9% normal saline Will be given as IV infusion Before anasthesia
  Interventions: Drug: placebo (100 mL of 0.9% saline).

INTERVENTIONS:
Drug: tranexamic acid (1 g diluted in 100 mL of 0.9% saline — The pharmacist also prepared indistinguishable infusion bags containing tranexamic acid (1 g diluted in 100 mL of 0.9% saline) . The infusion was administered intravenously over 10-15 minutes immediately after induction of anesthesia and before skin incision, at a maximum rate of 100 mg per minute
  Other Names: TXA
  Arms: tranexamic acid (1 g diluted in 100 mL of 0.9% saline
Drug: placebo (100 mL of 0.9% saline). — The pharmacist also prepared indistinguishable infusion bags containing placebo (100 mL of 0.9% saline). The infusion was administered intravenously over 10-15 minutes immediately after induction of anesthesia and before skin incision, at a maximum rate of 100 mg per minute
  Other Names: Inert saline
  Arms: placebo (100 mL of 0.9% saline).

SUMMARY:
Our study aims at evaluating the role of tranexamic acid in bariatric surgery since, The effect of conservative therapy using tranexamic acid for postoperative hemorrhage after bariatric surgery is still very much a novel technique. However,Intravenous tranexamic acid at the time of laparoscopic sleeve gastrectomy is associated with a significant reduction of post-operative bleeding with no observed differences in thromboembolic events or mortality.

DETAILED DESCRIPTION:
Participants were randomized in a 1:1 ratio to receive tranexamic acid or placebo using a computer-generated block randomization sequence (block size = 4) prepared by an independent pharmacist. Allocation concealment was maintained with sequentially numbered, opaque, sealed envelopes. The pharmacist also prepared indistinguishable infusion bags containing either tranexamic acid (1 g diluted in 100 mL of 0.9% saline) or placebo (100 mL of 0.9% saline). The infusion was administered intravenously over 10-15 minutes immediately after induction of anesthesia and before skin incision, at a maximum rate of 100 mg per minute. Blinding was maintained for patients, anesthesiologists, scrub nurses, and all postoperative assessors, while the operating surgeon was necessarily unblinded, becoming aware of allocation only once the envelope was opened in the operating room. All analyses were performed according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years were eligible if they had a body mass index (BMI) ≥ 35 kg/m², or ≥ 30 kg/m² with at least one obesity-related diseases(type 2 diabetes, hypertension, or obstructive sleep apnea).

Exclusion Criteria:

* Patients were excluded if they had a known coagulopathy or platelet disorder, a history of venous thromboembolism, myocardial infarction, or cerebrovascular accident, or if they on anticoagulant or antiplatelet therapy within ten days before surgery. Additional exclusion criteria included prior bariatric or major upper abdominal surgery, allergy or hypersensitivity to tranexamic acid, chronic kidney disease (stage 4-5), significant hepatic impairment, pregnancy or lactation.

Patient with alzheimer disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
intraoperative estimated blood loss (EBL | 10 DAYS
  Volume of blood loss in cm centimeter cubic
BLEEDING IN SLEEVE GASTRECTOMY | 10 DAYS
  Volume of blood loss in cubic centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Elshwadfy, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol: protocol only (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT07187258/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT07187258/SAP_001.pdf
  • Informed Consent Form (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT07187258/ICF_002.pdf